CLINICAL TRIAL: NCT03743870
Title: Spinal Anesthesia in Caesarean Section: Comparison Between Levobupivacaine and Hyperbaric Bupivacaine
Brief Title: Spinal Anesthesia in Caesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Collaborators: Marinella Astuto (Unknown)
Responsible Party: Principal Investigator, Carmelo Minardi, Principal Investigator, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Other Study IDs: 125/2018/PO
Record Dates: First submitted 2018-10-31; First posted 2018-11-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Hypotension Drug-Induced; Cesarean Section Complications; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use; Bradycardia
Keywords: intraoperative hypotension; bupivacaine; levobupivacaine; cesarean section; spinal anaesthesia; intraoperative bradycardia
MeSH Terms: conditions — Hypotension; Bradycardia | interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- levobupivacaine cohort: 125 pregnant patients that will have to undergo spinal anesthesia with Levobupivacaine for elective caesarean section.
  Interventions: Drug: Levobupivacaine
- bupivacaine cohort: Historical control group made of 125 patients underwent spinal anesthesia with Bupivacaine for elective cesarean section during the period between April 2017 and April 2018.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaine will be spinally administered, as required by normal clinical practice, at the dose of 12 mg 0,5% in combination with fentanyl 25γ.
  Groups: levobupivacaine cohort
Drug: Bupivacaine — Bupivacaine has been spinally administered, as required by normal clinical practice, at the dose of 12 mg 0,5% in combination with fentanyl 25γ.
  Groups: bupivacaine cohort

SUMMARY:
Spinal anesthesia is a safe technique, widely used and tested in the gynecological field, so as to be considered the first choice technique in cesarean section, which allows to quickly obtain a valid sensor and motor block. Bupivacaine is one of the most widely used drug for obtaining spinal anesthesia in pregnant women undergoing caesarean section. Bupivacaine is a local anesthetic available as a racemic mixture of its two enantiomers, the R (+)- dextrobupivacaine and the S (-) - levobupivacaine, whose clinical use is widely validated. Racemic bupivacaine is available as a simple or hyperbaric solution, the latter being the most commonly used for spinal anesthesia. Levobupivacaine, which is the pure levorotatory enantiomer of racemic bupivacaine, is a slightly hypobaric solution compared to liquor and has shown less heart and nerve toxicity, probably due to its ability to bind proteins more rapidly, and a greater selectivity towards the sensory component compared to Bupivacaine, presents action and effects better predictable. Its baricity would also offer the advantage of providing a less sensitive block to the position.

Hypotension is one of the most common complications of spinal anesthesia and is particularly relevant in caesarean section because, in addition to the adverse effects on the parturient, it can have repercussions on the fetus through a reduction of placental perfusion.

Some studies have showed a similar incidence of hypotension in patients treated with bupivacaine compared to those treated with levobupivacaine, while others assert an equivalence between the two drugs. In most studies, however, a significantly lower incidence of hypotension and a greater hemodynamic stability were reported in pregnant patients undergoing spinal anesthesia by caesarean section with levobupivacaine.

Being both hyperbaric bupivacaine and levobupivacaine routinely used at the "G. Rodolico" Universitary Hospital of Catania for the spinal anesthesia of pregnant women undergoing caesarean section and being their use decided exclusively at discretion of the treating anesthesiologist, in the light of the discrepant data in the literature about the incidence of hypotension with the two drugs, the main objective of this observational study is to evaluate the hemodynamic effects mediated by levobupivacaine on pregnant women subjected to elective cesarean section and to compare them with those mediated by hyperbaric bupivacaine in an historical court of pregnant women subjected to caesarean section in the period between April 2017 and April 2018. The hemodynamic parameters will be monitored in real time with a non-invasive hemodynamic monitoring system (EV1000® platform + Clearsight® system - Edwards LifeSciences), routinely used in the "G. Rodolico" Universitary Hospital of Catania, allowing to obtain greater accuracy and veracity of the results compared to previous studies conducted on such anesthetics.

DETAILED DESCRIPTION:
This is a prospective, monocentric, not for-profit, observational study, with historical control group, whose primary objective is the monitoring of changes in the hemodynamic condition, intended as continuous pressure measurements by means of a non-invasive system (EV1000® platform + Clearsight® system - Edwards Lifesciences), of a group of 125 pregnant women who have to undergo spinal anesthesia with Levobupivacaine for elective cesarean section at the "G. Rodolico" Presidium of Azienda Ospedaliero Universitaria "Policlinco-Vittorio Emanuele" of Catania, and to compare them with those detected, with the same non-invasive system, in an historical cohort of 125 patients who underwent spinal anesthesia with Bupivacaine for an elective caesarean section in the period between April 2017 and April 2018.

The study will have an expected duration of one year from the time of its approval.

In the levobupivacaine group, during the preoperative anesthesiological examination, carried out approximately two weeks before the scheduled date of the surgical intervention, informed consent will be acquired and the eligible patients will be enrolled. On this occasion, an ASA class will be assigned and the following data will be collected:

* personal and general data:

  * date of birth and age
  * current weight
  * weight before pregnancy
  * height
* information concerning:

  * any previous or concomitant diseases affecting the nervous, respiratory, cardiovascular system
  * any previous or concomitant disease interesting: gastrointestinal system, hemolymphatic system, thyroid, pancreas, kidneys, liver, adrenal glands
  * any immunodeficiencies
  * any coagulopathies
  * spinal deformities
  * previous surgeries
  * previous allergic events following the administration of drugs
  * seasonal allergies
  * previous pregnancies and their characteristics
  * possible hypertension during the last quarter
  * conditions that represent contraindications for spinal anesthesia. Upon arrival in the operating room, the Clearsight® non-invasive hemodynamic monitoring system will be placed at the fingers of the parturient and the usual intraoperative monitoring (ECG, non-invasive blood pressure, oxygen saturation) will be applied. The continuous recording of the following hemodynamic parameters, which will last for the whole duration of the intervention, will then begin through the EV1000® platform (Edwards Lifesciences): Cardiac Output (CO); Cardiac Index (CI); Stroke Volume (SV); Stroke Volume Index (SVI); Stroke Volume Variation (SVV); Pulse Rate Variation (PRV); Systemic Vascular Resistance (SVR); Systemic Vascular Resistance Index (SVRI); Central Venous Oxygen Saturation (ScvO2); Pulse rate (PR); Systolic Pressure (SYS); Diastolic Pressure (DIA); Mean Arterial Pressure (MAP); Central Venous Pressure (CVP).These measurements will be made every twenty seconds.

Once the monitoring system has been applied, the patients will be placed in position and spinal anesthesia will be performed with Levobupivacaine 12 mg 0.5% and Fentanyl 25γ. Once the anesthetic is injected, patients will be subjected to dislocation of the uterus and placed in left lateral tilt. Once the sensory and motor block has been obtained, the surgery will begin. In the event of adverse reactions to the drug, therapeutic measures that are part of the usual clinical practice will be used.

Any episodes of hypotension during the operation will be treated by administration of 5 mg etilefrine in bolus and/or IV fluids; any episodes of bradycardia will be treated by administration of IV atropine 0.01 mg/kg.

Sensory block will be evaluated by objective examination: the investigators will evaluate the tactile discrimination ability of a blunt tip in contact with the patient's back, thus determining the level of anesthesia reached and the time in which it occurs. The measurements of this parameter will be carried out every fifteen minutes, during the first half hour, and then at thirty and sixty minutes until the restitutio of the physiological condition of the patient.

The motor block will be evaluated by Bromage score, ie by observing the residual motor capacity of the patient's lower limbs. The measurements of this parameter will be carried out every fifteen minutes, during the first half hour, and then at thirty and sixty minutes until the restitutio of the physiological condition of the patient.

For calculating the Aldrete's score, the following parameters will be assessed: respiration and consciousness through objective examination, systolic blood pressure using the classic intraoperative monitoring system and pulse oximetry oxygenation. The measurements of this score will be carried out every fifteen minutes during the first half hour, and then at thirty and sixty minutes until the restitutio of the physiological condition of the patient.

Patient data from the historical cohort will be collected by reviewing the clinical documentation related to the individual case.

Once collected, the data will be subjected to statistical and comparative processing in order to highlight statistically relevant differences concerning the effects mediated by the two anesthetics on the pregnant patient who undergoes elective cesarean section.

The data obtained will be analyzed using the SPSS software (Statistical Package for Social Sciences), version 21.0 for Windows (SPSS Inc., Chicago, Illinois, USA). Differences with p≤ 0.05 will be considered significant.

The descriptive analysis will be performed using frequencies, percentages and frequency tables for qualitative variables. For the normally distributed quantitative variables the mean and standard deviation will be used, while for those not normally distributed the median and the interquartile range (IQR) will be used. For the comparison between the two groups will be used the Chi-square test with Yates correction or Fisher exact test for qualitative variables and the Mann-Whitney U test for quantitative variables.

Multivariate analysis will be performed using logistic regression models and the ORs (odds ratios) will be reported together with the corresponding 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* signature of informed consent
* age between 18 and 40 years old
* indication for spinal anesthesia
* American Society of Anesthesiology (ASA) classification I or II
* height less than 180 cm
* weight less than 100 kg
* absence of spinal deformities

Exclusion Criteria:

* age under 18 years old or over 40 yers old
* ASA III or IV
* contraindications to spinal anesthesia
* presence of hemodynamically relevant cardiovascular co-morbidities
* co-morbidities requiring invasive monitoring
* refusal of pregnant women to sign informed consent
* refusal of pregnant women to spinal anesthesia
* spinal deformities in pregnant women
* known hypersensitivity to the anesthetics used
* weight over 100 kg
* height over 180 cm
* preeclampsia or eclampsia
* presence of fetal or placental abnormalities such as placenta previa or placental abruption

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The study will involve consecutive pregnant womento to be subjected/subjected to spinal anesthesia for cesarean section at the Obstetric Emergency Room of the "G. Rodolico" Presidium of the Azienda Ospedaliero Universitaria "Policlinco-Vittorio Emanuele" of Catania that meet the inclusion and criteria of the study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in blood pressure measured continuously by the EV1000® platform and the Clearsight® non-invasive system (Edwards Lifesciences) in the two study cohorts | From arrival in the operating room until the completion of surgical procedures

SECONDARY OUTCOMES:
Incidence of hypotension during spinal anesthesia | At 60 minutes after completion of surgical procedures
Incidence of bradycardia during spinal anesthesia | At 60 minutes after completion of surgical procedures
Need for inotropes and / or vasopressor during surgery | At 60 minutes after completion of surgical procedures
  Doses of inotropes and / or vasopressor administered during surgery
Need for fluids administration during surgery | At 60 minutes after completion of surgical procedures
  Volume of fluids administered during surgery for the eventual treatment of hypotension
Level of the sensory block reached | At 15 minutes from the beginning of anesthesia
Time in which sensory block occurs | At 15 minutes from the beginning of anesthesia
Level of the sensory block reached | At 30 minutes from the beginning of anesthesia
Time in which sensory block occurs | At 30 minutes from the beginning of anesthesia
Level of sensory block reached | At 60 minutes from the beginning of anesthesia
Time in which sensory block occurs | At 60 minutes from the beginning of anesthesia
Level of the motor block reached by modified Bromage scale | At 15 minutes from the beginning of anesthesia
  The modified Bromage scale is a six-point scale used to asses the intensity of motor block by evaluation of the patient's ability to move their lower extremities: Score 1 = Complete block (unable to move feet or knees); Score 2 = Almost complete block (able to move feet only); Score 3 = Partial block (just able to move knees); Score 4 = Detectable weakness of hip flexion while supine (full flexion of knees); Score 5 = No detectable weakness of hip flexion while supine; Score 6 = Able to perform partial knee bend. The motor block is measured in both legs intermittently throughout labour, as the degree of block can change.
Level of the motor block reached by modified Bromage scale | At 30 minutes from the beginning of anesthesia
  The modified Bromage scale is a six-point scale used to asses the intensity of motor block by evaluation of the patient's ability to move their lower extremities: Score 1 = Complete block (unable to move feet or knees); Score 2 = Almost complete block (able to move feet only); Score 3 = Partial block (just able to move knees); Score 4 = Detectable weakness of hip flexion while supine (full flexion of knees); Score 5 = No detectable weakness of hip flexion while supine; Score 6 = Able to perform partial knee bend. The motor block is measured in both legs intermittently throughout labour, as the degree of block can change.
Level of the motor block reached by modified Bromage scale | At 60 minutes from the beginning of anesthesia
  The modified Bromage scale is a six-point scale used to asses the intensity of motor block by evaluation of the patient's ability to move their lower extremities: Score 1 = Complete block (unable to move feet or knees); Score 2 = Almost complete block (able to move feet only); Score 3 = Partial block (just able to move knees); Score 4 = Detectable weakness of hip flexion while supine (full flexion of knees); Score 5 = No detectable weakness of hip flexion while supine; Score 6 = Able to perform partial knee bend. The motor block is measured in both legs intermittently throughout labour, as the degree of block can change.
Aldrete score evaluation. | At 15 minutes from the beginning of anesthesia
  The evaluation of Aldrete score, also known Post Anesthesia Recovery (PAR), focuses on the following directions: muscle activity, assessed by observing the patient's ability to move his extremities on command; respiratory efficiency, reflected by the respiratory effort; circulation, evaluated through systemic blood pressure and compared to the preanesthetic level; consciousness, reflected by full alertness and ability to answer questions; tegument color, that evaluates whether the skin aspect is normal or cyanotic or jaundiced. Each of the five items in the Aldrete score calculation is awarded from 0 to 2 points, depending on the answer chosen in the evaluation. The higher the score, the more likelihood of recovery without need of observation. Results vary between 0 and 10. Patients with scores of 9 and 10 can be safely discharged from operatory room. Scores of 10 indicate a patient in the best condition. Scores of 7 and below come with indication of continuous close observation.
Aldrete's score evaluation | At 30 minutes from the beginning of anesthesia
  The evaluation of Aldrete score, also known Post Anesthesia Recovery (PAR), focuses on the following directions: muscle activity, assessed by observing the patient's ability to move his extremities on command; respiratory efficiency, reflected by the respiratory effort; circulation, evaluated through systemic blood pressure and compared to the preanesthetic level; consciousness, reflected by full alertness and ability to answer questions; tegument color, that evaluates whether the skin aspect is normal or cyanotic or jaundiced. Each of the five items in the Aldrete score calculation is awarded from 0 to 2 points, depending on the answer chosen in the evaluation. The higher the score, the more likelihood of recovery without need of observation. Results vary between 0 and 10. Patients with scores of 9 and 10 can be safely discharged from operatory room. Scores of 10 indicate a patient in the best condition. Scores of 7 and below come with indication of continuous close observation.
Aldrete's score evaluation | At 60 minutes from the beginning of anesthesia
  The evaluation of Aldrete score, also known Post Anesthesia Recovery (PAR), focuses on the following directions: muscle activity, assessed by observing the patient's ability to move his extremities on command; respiratory efficiency, reflected by the respiratory effort; circulation, evaluated through systemic blood pressure and compared to the preanesthetic level; consciousness, reflected by full alertness and ability to answer questions; tegument color, that evaluates whether the skin aspect is normal or cyanotic or jaundiced. Each of the five items in the Aldrete score calculation is awarded from 0 to 2 points, depending on the answer chosen in the evaluation. The higher the score, the more likelihood of recovery without need of observation. Results vary between 0 and 10. Patients with scores of 9 and 10 can be safely discharged from operatory room. Scores of 10 indicate a patient in the best condition. Scores of 7 and below come with indication of continuous close observation.

CONTACTS AND LOCATIONS:
Locations (1):
- "G. Rodolico" Presidium of the Azienda Ospedaliero Universitaria "Policlinico-Vittorio Emanuele", Catania, Italy